CLINICAL TRIAL: NCT04597775
Title: A Prospective, Randomized, Adaptive Phase II/III Clinical Trial, Controlled, Open-label, 3-arms, Parallel, Multi-centred, Chemoprevention of COVID-19: Hydroxychloroquine Post Exposure Prophylaxis For COVID-19
Brief Title: Chemoprevention Clinical Trial of COVID-19: Hydroxychloroquine Post Exposure Prophylaxis
Acronym: APCC-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Regional Center for Disease Control and Prevention, Jordan (Other)
Collaborators: Farhat Hached Hospital, Tunisia (Unknown); Fattouma Bourguiba, Tunisia (Unknown)
Responsible Party: Principal Investigator, Dr Munir Abu-Helalah, Chief Executive Officer, Regional Center for Disease Control and Prevention, Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APCC-19
Record Dates: First submitted 2020-10-18; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: SARS-CoV Infection
Keywords: COVID-19; SARS-CoV-2; Chemoprevention; Primary contact; Hydroxychloroquine; prophylaxis
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, open-label, three-arm, parallel, adaptive phase II/III controlled study in which subjects will be randomly assigned in a 1:1:1 ratio as per the following:
  Arm-1: hydroxychloroquine 800mg (400mg twice daily) given orally on day 1, (loading dose) hydroxychloroquine. Then 400mg (200mg 2 tablets) on day 2,3, 4 and 5.
  Arm-2: hydroxychloroquine 400mg (200mg twice daily) Given orally first day (loading dose), then 200mg once daily on day 2,3, 4 and 5.
  Arm-3: No Intervention- SARS-CoV-2 surveillance Standard control measures in the country of interest such as self isolation, good personal hygiene and good nutrition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 hydroxychloroquine 800mg day 1 and hydroxychloroquine 400mg day 2-5 (Experimental): hydroxychloroquine 800mg (400mg twice daily) given orally on day 1, (loading dose) hydroxychloroquine. Then 400mg (200mg 2 tablets) on day 2,3, 4 and 5.
  Interventions: Drug: hydroxychloroquine
- Arm 2 hydroxychloroquine 400mg day 1 and hydroxychloroquine 200mg day 2-5 (Active Comparator): hydroxychloroquine 400mg (200mg twice daily) Given orally first day (loading dose), then 200mg once daily on day 2,3, 4 and 5.
  Interventions: Drug: hydroxychloroquine
- No Intervention (No Intervention): No Intervention- SARS-CoV-2 surveillance Standard control measures in the country of interest such as self isolation, good personal hygiene and good nutrition.

INTERVENTIONS:
Drug: hydroxychloroquine — hydroxychloroquine
  Other Names: plaquenil
  Arms: Arm 1 hydroxychloroquine 800mg day 1 and hydroxychloroquine 400mg day 2-5; Arm 2 hydroxychloroquine 400mg day 1 and hydroxychloroquine 200mg day 2-5

SUMMARY:
Protocol summary

Title

A Prospective, randomized, adaptive phase II/III clinical trial, controlled, open-label, chemoprevention, 3-arms, parallel, multi-centred, to A Prospective, randomized, clinical trial, controlled, open-label, 3-arms, parallel, multi-centred, chemoprevention of COVID-19: Hydroxychloroquine Post Exposure Prophylaxis For COVID-19

Study Periods & Duration of Treatment

Study Duration: 6 months

Approval (IRB and regulatory bodies) 1 month

Recruitment and follow-up: 3 months

Analysis, report writing and submission of publications 1 month This study is a parallel study of one period with an expected duration of treatment (for each subject) of 28 days,

Objectives

* To evaluate if hydroxychloroquine with the proposed dose can provide potent chemoprophylaxis against the development of COVID-19 positive patients in subjects who had primary exposure to COVID-19 positive patients.
* To measure the incidence of potential adverse drug reaction rates for giving hydroxychloroquine for prevention of COVID-19 amongst close contacts
* To provide early analysis of results and redefine sample size accordingly.
* identifying subjects most likely to benefit during the phase II and focusing recruitment efforts on them during phase III
* stopping one arm or the whole trial at an early stage for success or lack of efficacy based on phase II study results

Design

Prospective, Randomized, open-label, three-arm, parallel, adaptive phase II/III controlled study in which subjects will be randomly assigned in a 1:1:1 ratio as per the following:

Arm-1: hydroxychloroquine 800mg (400mg twice daily) given orally on day 1, (loading dose) hydroxychloroquine. Then 400mg (200mg 2 tablets) on day 2,3, 4 and 5.

Arm-2: hydroxychloroquine 400mg (200mg twice daily) Given orally first day (loading dose), then 200mg once daily on day 2,3, 4 and 5.

Arm-3: No Intervention- SARS-CoV-2 surveillance Standard control measures in the country of interest such as self isolation, good personal hygiene and good nutrition.

DETAILED DESCRIPTION:
Type of study and design

Prospective, Randomized, open-label, three-arm, parallel, controlled adaptive phase II/III clinical trial in which subjects will be randomly assigned in a 1:1:1 ratio as per the following:

Arm 1 Arm 2 Arm 3 Day 1 HCQ 400 mg (twice daily) HCQ 200 mg (twice daily) Standard measurements of the country until the end of the participation in the study Day 2 HCQ 400 mg (once daily) HCQ 200 mg (once daily) Day 3 HCQ 400 mg (once daily) HCQ 200 mg (once daily) Day 4 HCQ 400 mg (once daily) HCQ 200 mg (once daily) Day 5 HCQ 400 mg (once daily) HCQ 200 mg (once daily)

Amount needed: Plaquenil 200mg: 558 tables per protocol. 42 tablets are needed as preserved supply: total 600 tables.

Randomisation Subjects who meet the eligibility criteria at the study locations will be invited to take part in the study.

Participants will be randomly assigned to the treatment arms. Index cases will be used for the assignment of contacts. For example, number 1,4,7, 9. will be on arm 1, number 3, 5, 10.etc. will be in arm 2, number 2,6, 8, etc. will be in arm 3.

All close contacts of the same index case will be allocated to the same arm. This would allow more valid results through prevention of potential further exposure to the virus mainly for the control arms, who are expected to have higher incidence of the disease.

Blinding This clinical trial is open-label. The study does not compare multiple medicinal products; it also does not include the use of a placebo product, as it is a Proamtic clinical trial.

Study procedures and evaluations Baseline assessment

* Medical history
* Inquiry about previous history of G6PD
* Check for contraindications
* Vital signs
* Physical examination
* RT-PCR
* IgM, IgG AB for SARS-Cov-2
* Hematology
* Biochemistry
* Urinalysis
* Retinopathy
* Pregnancy test
* ECG
* Retinopathy screening

During follow-up visits subjects will assessed for:

* Random glucose level
* Vital signs
* Assessment of study intervention adherence
* Assessment of adverse events.
* ECG
* Retinopathy screening Study schedule

Sampling technique:

This adaptive phase II/III clinical trial will be conducted in two sites in Tunisia. The main study is planned in 2 sites in Tunisia.

As soon as a new subject in identified, he/she will be consented for reaching his contacts according to Eligibility criteria. The research team within 48 hours of index case identification will call his/her contacts who fulfil below criteria for participation in the trial. All potential participants will be tested using RT-PCR and IgM and IgG antibodies to rule out current or previous disease status. Results will be obtained on the same day and before consenting for taking part in the study. Subjects positive for COVID-19 will be referred to local authorities for treatment according to their protocols.

We will follow multistage sampling technique in involved countries. Samples will be stratified by gender and then follow simple random sampling process.

Screening

Before carrying out any procedure in this study, subjects will be provided "subject information and consent form". The study will be thoroughly explained and all questions will be answered to the satisfaction of the subject. Subjects will be given enough time to think about their participation through and inquire about any detail that may influence the decision. Consent procedure will be carried out by the clinical investigator & delegated clinical staff. Neither the investigator nor the study staff will coerce or unduly influence subjects to participate or to continue to participate against their will. Prior to the subject's participation, the subject will personally sign & date the consent form, along with one witness at least & the principal investigator (the principal investigator may delegate the clinical investigator to sign the ICF whenever needed).

Enrollment (Baseline) All potential participants will be tested using RT-PCR and IgM and IgG antibodies to rule out current or previous disease status. Results will be obtained on the same day and before consenting for taking part in the study. Subjects positive for COVID-19 will be referred to local authorities for treatment according to their protocols.

Only subjects eligible for this study will be enrolled. Refer to section 5 for eligibility criteria.

Informed consent, , demographics, vital signs, Medical History and contraindications, physical examination,hematology, KFT, LFT, urinalysis,IgM and IgG antibodies for SARS-CoV-2, RT-PCR, Pregnancy test, ECG, Retinopathy screening, Blood Glucose, dosing, Adverse event review

During screening and follow-up visits, subjects will be examined and vital signs will be taken with relevant medical history taken to determine the lack of contraindication of the use the IMP and the achievement of the inclusion criteria Laboratory evaluations Laboratory evaluations will be conducted as per Table 6.1 of visits and procedures elaborated on table 6.1.

Safety considerations Methods and timing for assessing, recording, and analysing safety parameters Adverse events The study period during which adverse events must be reported is normally defined as the period from the initiation of any study procedures to the end of the study treatment follow-up. At each contact with the subject, the Clinical Investigator will seek information on adverse events by specific questioning and, as appropriate, by examination. Information on all adverse events will be recorded immediately in the source document, and also in the appropriate adverse event module of the case report form (CRF).

All adverse events occurring during the study period will be recorded. The clinical course of each event will be followed until resolution, stabilization, or until it has been determined that the study treatment or participation is not the cause. Serious adverse events that are still ongoing at the end of the study period will be followed up to determine the final outcome. Any serious adverse event that occurs after the study period and is considered to be possibly related to the study treatment or study participation should be recorded and reported immediately.

The AE report will include the intensity, severity, duration of the event. It will also explain how the case was managed. At the end of the study, all records and follow up forms of AEs/ADRs/SAEs/SADRs will be enlisted in the final report.

4 Discontinuation criteria 4.1 Participant's premature termination

The reason for participant's premature termination will be documented on the appropriate page of the CRF and specified which of the following possible reasons were responsible for the study premature termination:

* Serious Adverse Event / SUSAR
* Participant's consent withdrawal
* Inappropriate enrolment
* Development of exclusion criterion
* Protocol deviation: as described below:
* Such as not taking study treatment on time or the prescribed dose more than one time.
* Decline PCR test at baseline or during the follow-up
* Decline ECG or ophthalmoscopy exams.
* Migrated/moved from the study area
* Lost to follow-up. A 'lost to follow-up' is any participant who completed all protocol specific procedures up to the administration of the investigational product or intervention, but was then lost during the study period to any further follow-up, with no safety information and no efficacy endpoint data ever became available.

It is vital to collect safety data on any participant discontinued because of an AE or SAE. In any case, every effort must be made to undertake protocol-specified safety follow-up procedures. If voluntary withdrawal occurs, the participant should be asked to continue scheduled evaluations, complete an end-of-study evaluation, and be given appropriate care under medical supervision until the symptoms of any AE resolve or the participant's condition becomes stable.

5 Statistical considerations Following an adaptive seamless phase II/III design assuming 60% efficacy (an odds ratio of about 0.3) of hydroxychloroquine in reducing COVID-19 infections for primary contacts, and reported secondary attack rate of 35% (incidence amongst close contacts), Liu Y., et.al. 90% power, a confidence level of 95% and 10% loss to follow-up, 31 COVID-19 contacts are needed in each arm for phase II totaling 93 contacts for the three arms.

The primary endpoints of this study are observed COVID-19 infection and observed ADRs. Descriptive statistics including means, frequencies and proportions will be used to summarize collected contacts data. Incidence of the primary endpoints will be reported as well. All summaries will be provided for the three study arms. Chi-squared test will be used to compare incidence levels of the primary endpointsacross the three study arms. To examine for associations among categorical contacts attributes, Chi-squared and Fishers exact tests whenever appropriate will be used.When needed, ANOVA will be used to test for significant differences among numerical attributes.Logistic Regression techniques with stepwise selection method will be used to identify significant predictors of the primary endpoints Intention to treat analysis will be followed in this clinical trial

Data handling and record keeping Source documents and access to source data The Principal Investigators will maintain appropriate medical and research records for this study in compliance with the principles of good clinical practice and regulatory and institutional requirements for the protection of confidentiality of participants. The study team members will have access to records.

Authorised representatives of the sponsor, the ethics committee(s) or regulatory bodies may inspect all documents and records required to be maintained by the investigator for the purposes of quality assurance reviews, audits, inspections, and evaluation of the study safety and progress. This will include, but not limited to, medical records (office, clinic, or hospital) for the participants in this study. The clinical study site will permit access to such records.

Missing data will be reported as missing indicating the reasons where applicable.

Protocol deviations A protocol deviation is any noncompliance with the clinical trial protocol, good clinical practice (GCP), or other protocol-specific requirements.

If a deviation from, or a change of, the protocol is implemented to eliminate an immediate hazard(s) to trial participant without prior ethics approval, the PI or designee will submit the implemented deviation or change, the reasons for it, and, if appropriate, the proposed protocol amendment(s) as soon as possible to the relevant ethics committee(s) for review and approval and to the sponsor for agreement.

The PI or designee will document and explain any deviation from the approved protocol on the CRF, where appropriate, and record and explain any deviation in a file note or deviation form that will be maintained as an essential document.

Deviations from the protocol, GCP or trial specific requirements that might have an impact on the conduct of the trial or the safety of participants will be reported within 5 working days to the sponsor and relevant EC, as appropriate.

Ethical considerations The investigator will ensure that this study is conducted in full conformity with the principles set forth in the ICH Harmonised Tripartite Guideline for Good Clinical Practice and the Declaration of Helsinki in its current version, whichever affords the greater protection to the participants.

Rationale for participants election Study population will be males and females aged 18-65 years (non-pregnant and non-lactating) with primary exposure to COVID-19 patients. The study is proposed to be conducted in Tunisia.

Financing and insurance All subjects will be covered by insurance throughout the study and in case of an injury to health caused by the trial.

ELIGIBILITY:
Inclusion Criteria:

* Primary contacts, described below, aged 18 to 65 years and having provide Written informed consent by the patient, by the patient's legal /authorized representative as applicable.

According to below criteria, as soon as a new subject in identified, he/she will be consented for reaching his contacts according to below criteria. The research team within 48 hours of index case identification will call his/her contacts who fulfill below criteria for participation in the trial. All potential participants will be tested using RT-PCR and IgM and IgG antibodies to rule out current or previous disease status.

Contact is a person free from COVID-19 who experienced any one of the following exposures during the 2 days before and the 14 days after the onset of symptoms of a probable or confirmed case:

* A person living in the same household as a COVID-19 case
* A person having had direct physical contact with a COVID-19 case (e.g. shaking hands)
* A person having unprotected direct contact with infectious secretions of a COVID-19 case (e.g. being coughed on, touching used paper tissues with a bare hand)
* A person having had face-to-face contact with a COVID-19 case within 2 meters [2] and > 15 minutes
* A person who was in a closed environment (e.g. classroom, meeting room, hospital waiting room, etc.) with a COVID-19 case for 15 minutes or more and at a distance of less than 2 meters
* A healthcare worker (HCW) or other person providing direct care for a COVID-19 case, or laboratory workers handling specimens from a COVID-19 case without recommended personal protective equipment or with a possible breach of personal protective equipment use policies
* A contact in an aircraft sitting within two seats (in any direction) of the COVID-19 case, travel companions or persons providing care, and crew members serving in the section of the aircraft where the index case was seated (if severity of symptoms or movement of the case indicate more extensive exposure, passengers seated in the entire section or all passengers on the aircraft may be considered close contacts)

Exclusion Criteria:

* Women who are pregnant (at the time of screening) or breastfeeding
* known hypersensitivity or allergy to hydroxychloroquine or other aminoquinoline compounds
* History of severe skin reactions such as Stevens-Johnson syndrome and toxic epidermal necrolysis
* History of pre-existing retinopathy or maculopathy,
* concomitant use of tamoxifen
* History of congenital or acquired long QT-interval, current use of drugs that prolong the QT interval,
* family history of long QT arrythmia, cardiac disease such as heart failure, myocardial infarction
* concurrent use of anti-arrhythmic drugs, or family history of sudden cardiac death, or sudden cardiac death, bradycardia < 50 beats/min, uncorrected hypokalemia or hypomagnesemia
* severe renal disease or patients receiving dialysis
* Patients less than 35 kg bodyweight
* Currently taking Hydroxychloroquine
* Suspected or confirmed current COVID-19, defined as: (1) temperature > 38 Celsius; (2) cough; (3) shortness of breath; (4) sore throat; or, if available (not required), (5) positive confirmatory testing for COVID-19
* Inability to take medications orally
* Inability to provide written consent
* With significantly abnormal liver function
* Participants with psoriasis, myasthenia, hematopoietic and retinal diseases, CNS-related hearing loss;
* RT-PCR positive for SARS-CoV-2, IgM and IgG antibodies for SARS-CoV-2
* Currently using another treatment regimen or medication that is being investigated for efficacy in the management of COVID-19.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2020-10-27 (Estimated); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of COVID-19 on day 14 according to positive results of RT-PCR rate at day 14 | 14 days
  Study will seek to find direct correlation between the administration of Hydroxychloroquine and incidence of COVID-19: A reduced positive RT-PCR samples in subjects who were exposed to COVID-19patients. Positive RT-PCR samples in close contacts on day 14 of randomization.
Safety and adverse events (AEs) incidence rate at day 14 | 14 days
  Safety and adverse events (AEs) incidence rate at day 14

SECONDARY OUTCOMES:
IgM antibodies positive rate for COVID-19 at day 28 | 28 days
  Positive IgM antibodies
Incidence rate of COVID-19 on day 28 according to positive results of RT-PCR rate at day 28 | 28 days
  Positive at 28 days
Safety and adverse events (AEs) incidence rate on day 28 | 28 days
  Safety and adverse events (AEs) incidence rate on day 28

CONTACTS AND LOCATIONS:
Overall Officials: Munir Abu-Helalah, PHD, Principal Investigator — Regional Center for Disease Control; Wissem Hachfi, MD, Study Chair — Farhat Hached Hospital, Tunisia

IPD SHARING:
Plan to Share IPD: No
Through publications in Peer Review Journal